CLINICAL TRIAL: NCT01490099
Title: A Randomised, Single Centre, Double-blind, Two-period Cross-over Glucose Clamp Trial to Demonstrate Bioequivalence Between Insulin Detemir Produced by the NN729 Process and Insulin Detemir Produced by the Current Process in Healthy Subjects
Brief Title: Comparison of Insulin Detemir Produced by the Current Process and the NN729 Process in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX1729-1784; 2006-001677-17 (EudraCT Number)
Record Dates: First submitted 2011-12-06; First posted 2011-12-12 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Detemir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period 1 (Experimental)
  Interventions: Drug: insulin detemir
- Treatment period 2 (Active Comparator)
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — One single dose of insulin detemir produced by current process and the NN729 process injected subcutaneously on two separate dosing visits in varying order

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to demonstrate bioequivalence between insulin detemir produced by the NN729 process and by the current process in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history and physical examination as judged by the Investigator
* Body mass index (BMI) between 18.0 and 27.0 kg/m^2, inclusive
* Non-smoker
* Fasting plasma glucose (FPG) maximum 6.0 mmol/L

Exclusion Criteria:

* Known or suspected allergy to trial products or related products
* Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures (intrauterine device (IUD) that has been in place for at least 3 months, sterilisation, the oral contraceptive pill (which should have been taken without difficulty for at least 3 months) or an approved hormonal implant)
* A history of alcohol or drug abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2006-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
AUC0-36h, area under the serum insulin detemir concentration curve | From 0 to 36 hours
Cmax, maximum serum insulin detemir concentration

SECONDARY OUTCOMES:
AUC, area under the serum insulin detemir concentration curve
Time to maximum concentration (tmax)
Terminal half life (t½)
Area under the Curve Glucose Infusion Rate (AUCGIR)
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Manchester, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com